CLINICAL TRIAL: NCT01869777
Title: Investigating the Prognostic Importance of Bioelectrical Impedance Phase Angle in Adults Treated for Newly Diagnosed Acute Leukemia
Brief Title: Bioelectrical Impedance Measurement for Predicting Treatment Outcome in Patients With Newly Diagnosed Acute Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00023374; NCI-2013-00964 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 99113 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-05

CONDITIONS: Acute Undifferentiated Leukemia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Mast Cell Leukemia; Myeloid/NK-cell Acute Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Mast-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (bioelectric impedance analysis) (Experimental): Patients undergo bioelectrical impedance phase angle measurement on day 1 of treatment. Patients with AML undergo a second measurement just prior to the nadir marrow. Patients also undergo bioelectrical impedance measurements prior to any invasive procedures (bone marrow biopsy, leukapheresis, PICC line placement, etc.).
  Interventions: Procedure: bioelectric impedance analysis

INTERVENTIONS:
Procedure: bioelectric impedance analysis — Undergo bioelectric impedance analysis
  Other Names: BIA; bioelectric impedance; bioelectric impedance test; bioimpedance analysis

SUMMARY:
This clinical trial studies bioelectrical impedance measurement for predicting treatment outcome in patients with newly diagnosed acute leukemia. Diagnostic procedures, such as bioelectrical impedance measurement, may help predict a patient's response to treatment for acute leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I: To determine the feasibility of obtaining standardized phase angle measurements (bioelectrical impedance measurement) on patients hospitalized for treatment of newly diagnosed acute leukemia.

II. To evaluate the association between standardized phase angle measured at the start of therapy and treatment-related outcomes including treatment related mortality (defined as 60-day mortality) III. Evaluate the association of the day 14 standardized phase angle and treatment related outcomes, 30-day mortality, length of hospitalization, transfer to intensive care unit during induction, treatment response (14 day bone marrow response, complete remission), receipt of post-remission therapy, overall survival.

IV. An exploratory analysis investigating associations with the primary and secondary outcomes using different ways to categorize the baseline standardized phase angle and, for acute myeloid leukemia (AML) patients, the standardized phase angle measure obtained just prior to the nadir marrow.

OUTLINE:

Patients undergo bioelectrical impedance phase angle measurement on day 1 of treatment. Patients with AML undergo a second measurement prior to the nadir marrow. Patients also undergo bioelectrical impedance measurements prior to any invasive procedures (bone marrow biopsy, leukapheresis, peripherally inserted central catheter [PICC] line placement, etc.).

After completion of study treatment, patients are followed up for two years.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for newly diagnosed acute leukemia
* Receiving induction treatment while hospitalized
* Willing and able to provide written informed consent

Exclusion Criteria:

* Presence of a pacemaker or defibrillator
* Patients pregnant at the time of enrollment
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unable/unwilling to follow protocol requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pardee, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Started | 102
Completed | 101
Not Completed | 1
Not completed — Excluded from the analysis, ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Age, Continuous [Median (Full Range); unit: years] | 62.6 [22.9 to 83.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 91
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Treatment Related Mortality Defined as the Percent of Patients no Longer Alive at 60 Days After Registration
Description: Logistic regression will be used to analyze the association between standardized phase angle and 60 day mortality. 60 day mortality rate is defined as the percent of patients no longer alive at 60 days after registration. Patients that are discharged to hospice care before 60 days without a known date of death will be counted towards 60 day mortality
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Participants
  Alive | 91
  Deceased | 10

2. Secondary Outcome: Treatment Related Mortality Defined as the Percent of Patients no Longer Alive at 30 Days After Registration
Description: Logistic regression will be used to analyze the association between standardized phase angle and 30 day mortality. 30 day mortality rate is defined as the percent of patients no longer alive at 30 days after registration.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Participants
  Alive | 95
  Deceased | 6

3. Secondary Outcome: Length of Hospitalization
Description: A linear model will be used to look at the association of standardized phase angle and length of hospital stay.
Time Frame: Up to 2 years
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Days | 34.2 (11.9)

4. Secondary Outcome: Number of Participants Transferred to Intensive Care Unit During Induction
Description: Logistic regression will be used to analyze the association between standardized phase angle and transfer to intensive care unit.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Participants
  Transferred to ICU | 10
  Not transferred to ICU | 91

5. Secondary Outcome: Number of Participants With Bone Marrow Response
Description: Logistic regression will be used to analyze the significant association between standardized phase angle and marrow response at 14-day bone marrow biopsy to show the odds of having 14-day residual disease (presence cancer cells remaining after treatment) and non-residual disease (no cancer cells remaining after treatment). (14 day bone marrow response is defined as hypoplastic marrow with less than 20% cellularity and 5% blasts. Complete remission is defined as less than 5% marrow blasts, absolute neutrophil count >1000, platelet count >100,000 and freedom from red cell transfusions).
Time Frame: 14 days
Population: 14 participants excluded in analysis due to 14-day bone marrow data not available.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 87
Participants
  Residual disease | 47
  No residual disease | 40

6. Secondary Outcome: Number of Participants to Achieve Complete Remission
Description: Logistic regression will be used to analyze the association between standardized phase angle and complete remission. Complete remission is defined as less than 5% marrow blasts, absolute neutrophil count > 1000, platelet count > 100,000 and freedom from red cell transfusions
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Participants
  Achieved complete remission | 81
  Did not achieve complete remission | 20

7. Secondary Outcome: Number of Participants With Receipt of Post-Remission Therapy
Description: Logistic regression will be used to analyze the association between standardized phase angle and receipt of post-remission therapy.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Participants
  Receipt of post-remission therapy | 79
  Did not receive post-remission therapy | 22

8. Secondary Outcome: Overall Survival
Description: Association between overall survival and standardized phase angle will be evaluated using a Cox proportional hazards model.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
Number analyzed (Participants) | 101
Days | 532 [336 to 808]

ADVERSE EVENTS:
Time Frame: Up to 2 years to assess for survival only
Description: Adverse events were not monitored/assessed for this trial.
Arm/Group | Diagnostic (Bioelectric Impedance Analysis)
All-Cause Mortality (participants affected / at risk) | 16/101
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT01869777/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT01869777/ICF_002.pdf